CLINICAL TRIAL: NCT01076283
Title: A Pilot Study on the Biobehavioral Mechanisms of Baclofen and Alcohol Drinking
Brief Title: A Study on the Biobehavioral Mechanisms of Baclofen and Alcohol Drinking
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Lorenzo Leggio, Assistant Professor (Research), Brown University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0906000002
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Results first posted 2013-10-17 (Estimated); Last update posted 2013-10-17 (Estimated); Status verified 2013-10

CONDITIONS: Alcoholism
Keywords: baclofen; alcoholism; urge; craving; alcohol drinking; biobehavioral mechanisms of baclofen in alcoholism
MeSH Terms: conditions — Alcoholism; Alcohol Drinking | interventions — Baclofen; Cyproheptadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Baclofen (Active Comparator): Baclofen 10 mg three times a day (t.i.d.) for 8-10 days
  Interventions: Drug: Baclofen
- Cyproheptadine (Placebo Comparator): Cyproheptadine 2 mg t.i.d. for 8-10 days
  Interventions: Drug: Cyproheptadine

INTERVENTIONS:
Drug: Baclofen — Baclofen 10mg t.i.d.
  Arms: Baclofen
Drug: Cyproheptadine — 'active' placebo
  Arms: Cyproheptadine

SUMMARY:
This pilot trial has the goal to demonstrate the feasibility of a study to test the effects of baclofen in a laboratory experiment using cue-reactivity and alcohol-self administration paradigms in non-treatment seeking alcohol-dependent subjects.

ELIGIBILITY:
Inclusion Criteria:

* must be male or female between 21 and 65 years old (inclusive).
* participants must meet criteria for current Diagnostic and Statistical Manual of Mental Disorders, fourth edition, text revision (DSM-IV-TR) diagnosis of alcohol dependence, supported by the Structured Clinical Interview for DSM-IV-TR Axis I Disorders Patient Edition (SCID-I/P).
* participants must meet criteria for heavy drinking, defined as averaging ≥4 drinks/day for women and ≥5 drinks/day for men during a consecutive 30-day period within the 90 days prior to baseline evaluation (see: Anton et al, 2006). The gender-specific baseline was chosen as it represents heavy drinking that exceeds empirically based levels of moderate alcohol use that result in alcohol-related problems for women who consume ≥4 drinks/day, and men who consume ≥5 drinks/day (Sanchez-Craig et al, 1995).
* participants must be in good health as confirmed by medical history, physical examination, ECG, lab tests.
* females must be postmenopausal for at least one year, surgically sterile, or practicing an effective method of birth control before entry and throughout the study; have a negative urine pregnancy test at each visit.
* participants must be willing to take oral medication and adhere to the study procedures.

Exclusion criteria:

* individuals expressing interest in treatment for alcoholism.
* pregnancy or breast feeding women or not using an adequate form of birth control
* positive urine drug screen at baseline for any illegal substance (a urine drug screen may be repeated once during the screening period).
* individuals diagnosed with a current substance dependence diagnosis, other than alcohol or nicotine.
* meet DSM-IV Axis I criteria for a lifetime diagnosis of schizophrenia, bipolar disorder, or other psychoses.
* an active illness within the past 6 months of Visit 1 that meet the DSM-IV criteria for a diagnosis of Major Depressive Disorder (MDD) or Anxiety Disorder. Subjects with a history of suicide will be excluded.
* clinically significant medical abnormalities (i.e., unstable hypertension, ECG, bilirubin > 150% of the upper normal limit, ALT or AST elevations >300% the upper normal limit, creatinine clearance ≤ 60 dl/min).
* current use of psychotropic medications that cannot be discontinued that may have an effect on alcohol consumption or that may interact with baclofen or cyproheptadine.
* medical contraindications for use of baclofen or cyproheptadine.
* a history of adverse reaction or hypersensitivity to baclofen or cyproheptadine.
* individuals with a reasonable expectation of being institutionalized during the course of the trial.
* participants who have significant alcohol withdrawal symptoms, defined as a Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar) >10.
* history of seizures (e.g. epilepsy).
* subjects who have participated in any behavioral and/or pharmacological study within the past 90 days.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-12; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Leggio, M.D., M.Sc., Principal Investigator — Brown University Center for Alcohol and Addiction Studies
Locations (1):
- Brown University Center for Alcohol and Addiction Studies, Providence, Rhode Island, United States

REFERENCES:
- [Background] Leggio L, Garbutt JC, Addolorato G. Effectiveness and safety of baclofen in the treatment of alcohol dependent patients. CNS Neurol Disord Drug Targets. 2010 Mar;9(1):33-44. doi: 10.2174/187152710790966614. PMID 20201813
- [Background] Evans SM, Bisaga A. Acute interaction of baclofen in combination with alcohol in heavy social drinkers. Alcohol Clin Exp Res. 2009 Jan;33(1):19-30. doi: 10.1111/j.1530-0277.2008.00805.x. Epub 2008 Oct 6. PMID 18840257
- [Background] Addolorato G, Leggio L, Ferrulli A, Cardone S, Vonghia L, Mirijello A, Abenavoli L, D'Angelo C, Caputo F, Zambon A, Haber PS, Gasbarrini G. Effectiveness and safety of baclofen for maintenance of alcohol abstinence in alcohol-dependent patients with liver cirrhosis: randomised, double-blind controlled study. Lancet. 2007 Dec 8;370(9603):1915-22. doi: 10.1016/S0140-6736(07)61814-5. PMID 18068515
- [Background] Addolorato G, Leggio L, Abenavoli L, Agabio R, Caputo F, Capristo E, Colombo G, Gessa GL, Gasbarrini G. Baclofen in the treatment of alcohol withdrawal syndrome: a comparative study vs diazepam. Am J Med. 2006 Mar;119(3):276.e13-8. doi: 10.1016/j.amjmed.2005.08.042. PMID 16490478
- [Background] Addolorato G, Leggio L, Abenavoli L, DeLorenzi G, Parente A, Caputo F, Janiri L, Capristo E, Rapaccini GL, Gasbarrini G. Suppression of alcohol delirium tremens by baclofen administration: a case report. Clin Neuropharmacol. 2003 Sep-Oct;26(5):258-62. doi: 10.1097/00002826-200309000-00010. PMID 14520166
- [Background] Addolorato G, Leggio L, Abenavoli L, Caputo F, Gasbarrini G. Tolerance to baclofen's sedative effect in alcohol-addicted patients: no dissipation after a period of abstinence. Psychopharmacology (Berl). 2005 Mar;178(2-3):351-2. doi: 10.1007/s00213-004-2014-4. Epub 2004 Sep 30. No abstract available. PMID 15719231
- [Background] Colombo G, Addolorato G, Agabio R, Carai MA, Pibiri F, Serra S, Vacca G, Gessa GL. Role of GABA(B) receptor in alcohol dependence: reducing effect of baclofen on alcohol intake and alcohol motivational properties in rats and amelioration of alcohol withdrawal syndrome and alcohol craving in human alcoholics. Neurotox Res. 2004;6(5):403-14. doi: 10.1007/BF03033315. PMID 15545024
- [Background] Addolorato G, Caputo F, Capristo E, Domenicali M, Bernardi M, Janiri L, Agabio R, Colombo G, Gessa GL, Gasbarrini G. Baclofen efficacy in reducing alcohol craving and intake: a preliminary double-blind randomized controlled study. Alcohol Alcohol. 2002 Sep-Oct;37(5):504-8. doi: 10.1093/alcalc/37.5.504. PMID 12217947
- [Result] Leggio L, Zywiak WH, McGeary JE, Edwards S, Fricchione SR, Shoaff JR, Addolorato G, Swift RM, Kenna GA. A human laboratory pilot study with baclofen in alcoholic individuals. Pharmacol Biochem Behav. 2013 Feb;103(4):784-91. doi: 10.1016/j.pbb.2012.11.013. Epub 2012 Dec 19. PMID 23262301

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants came for an in-person screening (Visit 1) at the Brown University Center for Alcohol and Addiction Studies (CAAS). At Visit 2 (day 1), participants were randomized to either baclofen or active placebo by using a 3-urn variable procedure (Stout et al., 1994), i.e. gender, FH of alcoholism and baseline drinks per drinking day.
Pre-assignment Details: 19 participants signed the consent document; 5 of them did not satisfy the protocol-specific inclusion/exclusion criteria, therefore they were excluded from the trial. The remaining 14 subjects were assigned to the study groups.
Period: Overall Study
Arm/Group | Baclofen | Cyproheptadine
Started | 7 | 7
Completed | 6 | 7
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Baclofen | Cyproheptadine | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Urge
Description: Whether baclofen, as compared to active placebo, results in diminished cue-reactivity responses to alcohol cues in terms of urge to drink [as measured by the Alcohol Urge Questionnaire (AUQ)] during the Cue Reactivity.
  The Alcohol Urge Questionnaire (AUQ) consists of eight statements about the respondent's feelings and thoughts about drinking as they are completing the questionnaire (i.e., right now). The respondent is asked to respond to each statement about alcohol craving via a 7-item Likert scale ranging from "strongly disagree" to "strongly agree." Each item is scored on a 1 to 7 scale (Strongly Disagree = 1 and Strongly Agree = 7). Items 2 and 7 are reverse scored. A total score is computed by summing the item scores and ranges from 8 (lowest craving value) to 56 (highest craving value). Higher scores reflect greater craving (i.e. worse outcome).
Time Frame: approximately 8 days after drug administration
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baclofen | Cyproheptadine
Number analyzed (Participants) | 6 | 7
units on a scale | 22.5 (11.4) | 19.4 (19.6)

2. Primary Outcome: Alcohol Drinking
Description: Whether baclofen, as compared to active placebo, results in lower quantity of alcohol consumed during the Alcohol Self-Administration (ASA).
  Consistent with O'Malley et al. 2002, the ASA paradigm allows to use a fixed-dose (the priming drink), followed by a 2-hour "free-choice" phase when subjects may choose to drink or not up to 8 mini-drinks. Participants receive a monetary compensation of $3 dollars per each mini-drink not consumed; therefore the amount of minidrinks consumed during the 2-hour sessions ranges 0-8, and the monetary compensation ranges $0-24. The quantity of alcohol consumed during the free-choice session is expressed as "standard drinking unit", where a standard drink unit contains about 14 grams of pure alcohol (about 0.6 fluid ounces or 1.2 tablespoons).
Time Frame: approximately 8 days after drug administration
Measure: Mean (Standard Deviation); unit: standard drinking units
Arm/Group | Baclofen | Cyproheptadine
Number analyzed (Participants) | 6 | 7
standard drinking units | 0.17 (0.41) | 1.43 (2.30)

ADVERSE EVENTS:
Arm/Group | Baclofen | Cyproheptadine
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 6/7 | 3/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baclofen (N=7) | Cyproheptadine (N=7)
sleepness (Nervous system disorders) | 2 | 1
increased urination (Renal and urinary disorders) | 1 | 0
cramps (Musculoskeletal and connective tissue disorders) | 1 (2) | 0
constipation (Gastrointestinal disorders) | 0 | 1
yellow urine (Renal and urinary disorders) | 0 | 1
sedation (Nervous system disorders) | 3 | 2
diarrhea (Gastrointestinal disorders) | 1 | 0
loss of libido (Reproductive system and breast disorders) | 1 | 0
nausea (Gastrointestinal disorders) | 1 | 0
insomnia (Nervous system disorders) | 1 | 0
irritability (Nervous system disorders) | 1 | 0
flatulence (Gastrointestinal disorders) | 1 | 0
neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
dental pain (General disorders) | 0 | 1
stomachache (Gastrointestinal disorders) | 1 | 0
foggy (Nervous system disorders) | 1 | 0
'high' (Nervous system disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Very small sample. This pilot trial was primarily aimed to determine a power analysis for future larger trials.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes